CLINICAL TRIAL: NCT02188693
Title: Maintenance Versus Observation With 6 Cycles of Gemcitabine Plus Taxol Sequential Gemcitabine Single Agent in Patients With Metastatic Breast Cancer
Brief Title: Gemcitabine as a Single Agent in the Maintenance Chemotherapy of Patients With Metastatic Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, LiNanlin,Ph.D, Chief Physician,Clinical Professor, The department of Vascular endocrine surgery, Xijing Hospital
Other Study IDs: NLLY-01
Record Dates: First submitted 2014-07-09; First posted 2014-07-14 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Stage IIIB, IV, Recurrent, and Metastatic Breast Cancer; Gemcitabine; Maintenance Chemotherapy
MeSH Terms: conditions — Recurrence; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — 2 ml blood sample is needed before enrollment.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Gemcitabine, Experimental: Gemcitabine 1250 mg/m2, IV on day 1 of 21 day cycle,with a follow up for every 12 weeks until disease progression or the date of first documented death from any cause
- Observational: Observation for every 12 weeks until disease progression or the date of first documented death from any cause

SUMMARY:
The primary purpose of our study is to evaluate whether gemcitabine as a single agent is superior to observation in improving progression-free survival (PFS) in patients with metastatic breast cancer (MBC) who achieved disease control with an initial six cycles of PG as their first-line treatment

ELIGIBILITY:
Inclusion Criteria:

* Histologically Confirmed Metastatic, or Recurrent Breast Cancer
* Age over 18 Years
* ECOG Performance Status 0-2
* Premenopausal or Postmenopausal Breast Cancer Patients With Measurable or Non-Measurable Lesions, Who Are Candidates for Chemotherapy
* Life Expectancy ≥ 3 Months
* Patients May Have Received Prior Neoadjuvant or Adjuvant Taxane Regimen as Long as it Has Been 12 Months Since Completion of Regimen.
* Patients Either May or May Not Have a Prior Anthracycline Containing Regimen.
* Prior Hormonal Therapy as a Treatment of Metastatic Disease is Allowed. But Antitumoral Hormonal Therapy Must be Terminated Prior to Enrollment(up to the Date of Randomization)
* Prior Radiation Therapy Allowed as Long as < 25% of the Bone Marrow Has Been Treated,and the Patients Must Have Recovered From the Acute Toxic Effects of the Treatment Prior to Study Enrollment.Prior Radiation to the Whole Pelvis is Not Allowed. Prior Radiotherapy Must be Completed 4 Weeks Before Study Entry.
* Adequate Bone Marrow Function (≥ ANC 1,500/ul, ≥ Platelet 100,000/ul, ≥ Hemoglobin 9.0 g/dl)
* Adequate Renal Function (≤ Serum Creatinine 1.5 mg/dl or CCr ≥ 50 ml/Min)
* Adequate Liver Function (≤ Serum Bilirubin 1.5 mg/dl, ≤ AST/ALT x 3 Upper Normal Limit)
* No Prior History of Chemotherapy for Metastatic, Recurrent Breast Cancer
* Written Informed consent

Exclusion Criteria:

* Serious Uncontrolled Intercurrent Infections
* Serious Intercurrent Medical or Psychiatric Illness, Including Active Cardiac Disease
* Pregnancy or Breast Feeding
* Second Primary Malignancy(Except Cancer of Cervix or Skin or Other Malignancy Treated at Least 5 Years Previously With no Evidence of Recurrence)
* Documented Parenchymal or Leptomeningeal Brain Metastasis
* Peripheral Neuropathy ≥ Grade 2
* Prior Treatment With Gemcitabine Will Not be Allowed.
* HER-2 Overexpressing Breast Cancer and Concomitant Trastuzumab Treatment is Not Allowed

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with MBC exhibited disease control (complete response + partial response + stable disease) with first-line PG and were randomly assigned to maintenance chemotherapy or observation.
Sampling Method: Non-Probability Sample
Enrollment: 267 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
PFS | From randomization to disease progression
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
PFS(progression free survival) | time from the date of randomization until the date of disease progression，assessed up to 3 years
PFS(progression free survival) | the time from the date of randomization until the date of disease progression,assessed up to 3 years
  PFS was defined as the time from the date of randomization until the date of disease progression at any site including distant metastasis or second primary tumors or death,assessed up to 3 years

SECONDARY OUTCOMES:
OS(overall survival) | the time from date of randomization until the date of first documented death from any cause,assessed up to 3 years
  the time from date of randomization until the date of first documented death from any cause,assessed up to 3 years

OTHER OUTCOMES:
QoL(quality of life) | the time from enrollment to disease progression or the date of first documented death,assessed up to 3 years
  the time from enrollment to disease progression or the date of first documented death,whichever comes first,to observe the quality of life in participants,assessed up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Li Nanlin, Ph.D, Study Director — Air Force Military Medical University, China
Locations (1):
- Xijing Hospital ， Fourth Military Medical University, Xi'an, Shaanxi, China